CLINICAL TRIAL: NCT00404209
Title: Pressurized Perfluorocarbon Perfused 23 GA Vitrectomy in Complicated Diabetic Retinal Detachment
Brief Title: Pressurized PPV 23GA Vitrectomy in Complicated Diabetic Tractional Retinal Detachment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Hugo Quiroz-Mercado, Asociacion para evitar la ceguera en Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-008
Record Dates: First submitted 2006-06-30; First posted 2006-11-28 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — pressurized 23GA vitrectomy with a 3D system

SUMMARY:
To investigate the feasibility and advantages of using pressurized perfluorocarbon liquid (PCL) perfusion to remove vitreous during suction-cutting 23 GA vitrectomy using a dual, dynamic drive (3D)technology, in complicated retinal detachment surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Complicated retinal detachment with no more than 6months of evolution

Exclusion Criteria:

* Retinal detachments of more than 6 months of evolution No light perception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Perfluorocarbon liquids consumption | two months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico, Hospital "Luis Sanchez Bulnes"; Raul Velez-Montoya, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México, Hospital "Luis Sánchez Bulnes", Mexico City, Mexico DF, Mexico